CLINICAL TRIAL: NCT00972400
Title: Biological Mechanisms of Fatigue in Breast Cancer Survivors
Brief Title: Fatigue in Breast Cancer Survivors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St George's, University of London (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000647658; SGUL-PTF-Mechanisms; EU-20958
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2009-09

CONDITIONS: Breast Cancer; Cancer Survivor; Fatigue; Psychosocial Effects of Cancer and Its Treatment
Keywords: psychosocial effects of cancer and its treatment; fatigue; cancer survivor; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Fatigue | interventions — Mass Spectrometry; Mental Status and Dementia Tests

INTERVENTIONS:
Genetic: protein analysis
Other: laboratory biomarker analysis
Other: mass spectrometry
Other: questionnaire administration
Procedure: assessment of therapy complications
Procedure: cognitive assessment
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Gathering information over time from blood samples and measurements of activity, sleep, mood, and cognition may help doctors learn more about fatigue in breast cancer survivors and plan the best treatment.

PURPOSE: This clinical trial is studying fatigue in breast cancer survivors.

DETAILED DESCRIPTION:
OBJECTIVES:

* To investigate the relationship between fatigue severity; protein biomarkers; and measures of activity, sleep, mood, and cognition in breast cancer survivors.
* To identify and quantify serum biomarkers and underlying biological pathways unique to cancer-related fatigue syndrome in these survivors.
* To map changes over time in order to explore the inter-relationships between these variables.

OUTLINE: Participants undergo fatigue assessment by the Diagnostic Interview for Cancer Related Fatigue and the FACT-Fatigue questionnaire; psychological symptoms assessment by the Structured Clinical Interview for DSM-IV, Hospital Anxiety and Depression Scale, and the Insomnia Severity Index questionnaires; and quality of life assessment by the EORTC-QLQc30 and EORTC-QLQ-BR23 questionnaires twice approximately 3 months apart.

Participants also undergo activity level, circadian rhythm, and sleep measurements by the Micro-mini® Motionlogger actigraphy and measurement of cognitive disturbances by the Cantabeclipse™ technology.

Participants undergo blood sample collection for protein analysis by 2D gel electrophoresis and mass spectrometry.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Disease-free breast cancer survivors between 3 months and 2 years after completion of primary treatment
* Recruited from the nurse-led breast cancer follow-up clinic at St George's Hospital

PATIENT CHARACTERISTICS:

* Sufficient English language skills
* No significant cognitive impairment
* No concurrent severe combined immunodeficiency disease

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Relationship between fatigue severity; protein biomarkers; and measures of activity, sleep, mood, and cognition
Identification and quantification of serum biomarkers underlying biological pathways unique to cancer-related fatigue syndrome
Inter-relationships between variables

CONTACTS AND LOCATIONS:
Overall Officials: Ollie Minton, MD, Principal Investigator — St George's, University of London
Locations (1):
- St. Georges, University of London, London, England, United Kingdom